CLINICAL TRIAL: NCT07162571
Title: Phase I/II Open-label Study Evaluating The Safety And Efficacy of Anti CD19/22 CAR-T Cells Therapy Adults With R/ R Leukemia/ Lymphoma
Brief Title: This is a Phase I/II Interventional, Open-label Treatment Study Designed to Evaluate the Safety and Efficacy of Anti CD 19/22 CAR- T Cells Immunotherapy for Adults With Relapsed or Refractory Acute Lymphoblastic Leukemia/Lymphoma.
Acronym: MSTH-CAR002
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Minsk Scientific-Practical Center for Surgery, Transplantation and Hematology (Other Government)
Responsible Party: Principal Investigator, Mikhail Uss, Dr. Mikhail Uss. Head of the Department of Bone Marrow Transplantation, Researcher, Minsk Scientific-Practical Center for Surgery, Transplantation and Hematology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23.25
Record Dates: First submitted 2025-08-29; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Acute Lymphobkastic Leukemia; B Cell Lymphoma
Keywords: CD19/22 CAR-T cells; Acute Lymphobkastic Leukemia; B Cell lymphoma; dual targeting CAR-T therapy
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19/22 CAR-T cells immunotherapy (Experimental)
  Interventions: Biological: CD19/22 CAR-T cells

INTERVENTIONS:
Biological: CD19/22 CAR-T cells — Following preconditioning with chemotherapy (cyclophosphamide and fludarabine) patients will be treated with doses from 50 x 10⁶ to 150 x 10⁶ CD19/CD22 CAR-T cells

SUMMARY:
The purpose of this study is to estimate the safety and the efficacy of anti-CD19/22 CAR- T cells immunotherapy for adults with relapsed or refractory acute lymphoblastic leukemia/lymphoma.

DETAILED DESCRIPTION:
Locally manufactured second generation autologous CD19/22 CAR-T cells are used for immunotherapy. Protocol treatment includes leukapheresis in order to harvest T cells, lymphodepleting conditioning (fludarabine + cyclophosphamide) followed by one dual targeting CAR-T cells infusion.

The Main research objectives of the Phase I:

To preliminarily explore the safety (incidence of CRS, ICANS, HLH, infections, late ICAHT, and cytopenias) and tolerability.

The Secondary research objectives of the Phase I:

To explore the pharmacokinetics of CAR-T cells.

The Main research objectives of the Phase II:

Overall response rate, including complete response (CR) and partial response (PR) rates.

The Secondary research objectives of the Phase II:

Duration of response (DOR). Progression-free survival rates. Overall survival rates.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥18 years.
2. Willing and able to give written, informed consent.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 1.
4. Relapsed or refractory lymphoblastic leukemia/lymphoma.

   - Chemotherapy-refractory disease after ≥1 lines of therapy

   - Relapse after chemotherapy or after ASCT/Allo-HSCT.
5. Adequate organ system function including - Creatinine clearance ≥40 cc/min.

   - Serum alanine aminotransferase / aspartate aminotransferase ≤2.5 x upper limit of normal (ULN).

   - Total bilirubin ≤1.5 x ULN, except in subjects with Gilbert's syndrome.

   - Left ventricular ejection fraction (LVEF) ≥50% (by echocardiogram [ECHO] or

   - Baseline oxygen saturation >92% on room air and ≤Grade 1 dyspnoea.
6. Have no active GVHD (Grade 2-4)
7. Adequate bone marrow (BM) function - Absolute neutrophil count ≥1.0 × 10^9/L.

   * Absolute lymphocyte count ≥0.3 × 10^9/L (at enrolment and prior to leukapheresis).
   * Haemoglobin ≥80 g/L.
   * Platelets ≥75 × 10^9/L

7. The expression of CD19 and/or CD22 on the tumor cells are reported as positive by either immunohistochemistry or flow cytometry

Exclusion Criteria:

1. Females who are pregnant or lactating.
2. History or presence of clinically relevant CNS pathology such as epilepsy, paresis, aphasia, stroke within prior 3 months, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, uncontrolled mental illness, or psychosis.
3. Patients with active CNS involvement by malignancy. Patients with history of central nervous system (CNS) involvement with malignancy may be eligible if CNS disease has been effectively treated and provided treatment was at least 4 weeks prior to enrolment (at least 8 weeks prior to CAR-T infusion).
4. Clinically significant, uncontrolled heart disease or a recent (within 12 months) cardiac event.
5. Active bacterial, viral or fungal infection requiring systemic treatment. Active or latent hepatitis B infection or hepatitis C infection. Testing positive for human immunodeficiency virus, human T cell lymphotropic virus (HTLV1 and 2) or syphilis.
6. History of autoimmune disease resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 24 months.

6. Evidence of active pneumonitis on chest computed tomography (CT) scan at screening or history of drug-induced pneumonitis, idiopathic pulmonary fibrosis, organising pneumonia, or idiopathic pneumonitis.

7. History of other malignant neoplasms unless disease free for at least 24 months (carcinoma in situ, non-melanoma skin cancer, breast or prostate cancer on hormonal therapy allowed).

8. The following medications are excluded:

* Steroids: Therapeutic doses of corticosteroids within 7 days of leukapheresis or 72 hours prior to CAR-T administration. However, physiological replacement, topical, and inhaled steroids are permitted.
* Immunosuppression: Immunosuppressive medication must be stopped ≥2 weeks prior to leukapheresis or CAR-T cells infusion.
* Cytotoxic chemotherapies within 1 week of CAR-T cellsinfusion and 1 week prior to leukapheresis.
* Antibody therapy use including anti-CD20/19/22 therapy within 2 weeks prior to CAR-T cells infusion.
* Granulocyte-colony stimulating factor less than 14 days prior to leukapheresis.
* Live vaccine ≤4 weeks prior to enrolment.
* Prophylactic intrathecal therapy: Methotrexate within 4 weeks and other intrathecal chemotherapy (e.g. Ara-C) within 2 weeks prior to starting pre-conditioning chemotherapy.

Prior limited radiation therapy within 2 weeks of CAR-T cells infusion. 9. Known allergy to albumin, dimethyl sulphoxide (DMSO), cyclophosphamide or fludarabine or tocilizumab.

10. Any other condition that in the Investigator's opinion would make the patient unsuitable for the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Phase I. Safety | 1 month post CAR-T cells infusion
  Number of Participants With Grade 3-5 Toxicities. Adverse events will be graded according to the CTCAE v5.0
Phase II. Overall response rate | 3 months post CAR-T cells infusion
  Including complete response (CR) and partial response (PR) rates

SECONDARY OUTCOMES:
Phase I. CAR-T proliferation | 3 months post CAR-T cells infusion
  To explore the pharmacokinetics of CAR-T cells: duration of expansion of CAR-T cells by flow cytometry, peak of expansion of CAR-T cells
Phase II. Efficacy: Overall survival rates | 12 months post CAR-T cells infusion
  Overall survival rates
Phase II. Progression-free survival rates | 12 months post CAR-T cells infusion
  progression-free survival time
Phase II. Duration of response | 12 months post CAR-T cells infusion
  duration of response

CONTACTS AND LOCATIONS:
Locations (1):
- State Institution Minsk Scientific and Practical Center for Surgery, Transplantology, and Dermatology, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR